CLINICAL TRIAL: NCT04946929
Title: Determine the Safety/Efficacy of Ticagrelor in Post-transplant Patients With Hepatic Artery Thrombosis (HAT)
Brief Title: Ticagrelor in Post-transplant Patients With Pediatric Hepatic Artery Thrombosis (HAT)
Acronym: Tip-HAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2021-083
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Hepatic Artery Thrombosis; Liver Transplant; Complications; Pediatric Disease
MeSH Terms: interventions — Ticagrelor; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ticagrelor, 2-3mg/kg, 12h (Experimental): 2-3mg/kg, q12h, p.o. for 2w
  Interventions: Drug: Ticagrelor Oral Tablet [Brilinta]
- low molecular weight heparin (Active Comparator): half amount low molecular weight heparin
  Interventions: Drug: Low molecular weight heparin

INTERVENTIONS:
Drug: Ticagrelor Oral Tablet [Brilinta] — Ticagrelor, 2-3mg/kg, 12h, p.o.
  Other Names: Ticagrelor
  Arms: Ticagrelor, 2-3mg/kg, 12h
Drug: Low molecular weight heparin — half amount low molecular weight heparin
  Arms: low molecular weight heparin

SUMMARY:
Hepatic artery thrombosis (HAT) represents a major cause of graft loss and mortality after Pediatric liver transplantation. Ticagrelor (a new reversible inhibitor of P2Y12 receptor with faster onset of action and greater platelet inhibition) was used to treat patients with pediatric post-transplant hepatic artery thrombosis (HAT) compared to low molecular weight heparin.

DETAILED DESCRIPTION:
In pediatric patients with post-transplant hepatic artery thrombosis (HAT) , low molecular weight heparin is a commonly used method. Ticagrelor, a direct-acting and reversible ADP receptor antagonist, is now the most commonly used ADP receptor antagonist in the treatment of coronary diseases. Compared to its predecessor clopidogrel, the pharmacokinetic profil of ticagrelor is more predictable, demonstrating a faster onset of action and a more consistent platelet inhibition. However, because of the excellent antithrombotic effect and increased bleeding potential, it is recommended that major bleeding, such as OPCAB or CABG surgery, be expected with a high probability, and in case of fatal surgery, the drug should be discontinued for 5 days. The present study is to evaluate the safety and efficacy of Ticagrelor in pediatirc receipt with post-operative HAT.

ELIGIBILITY:
Inclusion Criteria:

* age from 2 months to 5 years old.
* voluntary participation in clinical trials, and informed consent;
* Contrast- Enhanced Ultrasonography proved HAT

Exclusion Criteria:

* History of sensitivity to study medications or any of their excipients
* Renal failure (eGFR <30 or requiring dialysis)
* A known bleeding diathesis, hemostatic or coagulation disorder, or prior major bleeding
* Prior stroke
* Active pathological bleeding
* History of intracranial haemorrhage
* Life expectancy <12 months based on investigator's judgement
* Patients considered to be at risk of bradycardic events (e.g., known sick sinus syndrome or second or third degree atrioventricular [AV)] block) unless already treated with a permanent pacemaker
* Anemia (hematocrit < 27%)
* Platelet count < 100,000/ml
* Concomitant use of strong CYP 3A inhibitors or inducers

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Contrast-Enhanced Ultrasonography-Based Hepatic Perfusion Index | 3 months
  The peak systolic maximum velocity (Vmax) of the HA, and HA resistive index (HARI)

SECONDARY OUTCOMES:
High on-treatment platelet reactivity (HPR) | Two hours after the injection of either active drug or placebo
  HPR defined as platelet reactivity index (PRI) ≥50% using VASP analysis
Post-operative major bleeding event | within 72 hours after operation
  post-operative major bleeding defined as HAT related bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Hao Feng, MD. Ph.D, Principal Investigator — Dept. Liver Surgery, Renji Hospital affiliated to Shanghai Jiao Tong University School of Medicine; Chuan Shen, MD, Principal Investigator — Dept. Liver Surgery, Renji Hospital affiliated to Shanghai Jiao Tong University School of Medicine; Xiaosong Chen, MD, Study Director — Dept. Liver Surgery, Renji Hospital affiliated to Shanghai Jiao Tong University School of Medicine; Qiang XIA, MD. Ph.D, Study Chair — Dept. Liver Surgery, Renji Hospital affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China